CLINICAL TRIAL: NCT00516178
Title: Effects of Intravenous n-3 Polyunsaturated Fatty Acid Administration in Critically Ill Cardiac Surgery and Myocardial Infarction Patients
Brief Title: Intravenous Fish Oil in Critically Ill Cardiac Patients
Acronym: FO-cardiac
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Mette M Berger, Prof, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FN-3200BO-102064
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease
Keywords: Fish oil supplement; n-3 PUFA; Cardiac function; Membrane incorporation; Inflammation; Clinical outcome
MeSH Terms: conditions — Coronary Artery Disease; Inflammation | interventions — fish oil triglycerides; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Saline (No lipid emulsion)
  Interventions: Drug: Saline
- Fish oil emulsion (Experimental): 3 infusions of 0.2 g/kg omega-3 PUFA within 24 hours in cardiac surgery (continuous infusion post-PTCA)
  Interventions: Drug: Fish oil emulsion

INTERVENTIONS:
Drug: Fish oil emulsion — 0.2 g/kg FO, 3 times in 24 hours, infused over 3 hours each in cardiac surgery, or continuous infusion of 0.6 g/kg post PTCA
  Other Names: Omegaven,Fresenius Kabi AG
  Arms: Fish oil emulsion
Drug: Saline — 3 infusions, perioperative or post-PTCA
  Arms: Placebo

SUMMARY:
A large body of evidence has accumulated showing that n-3 PUFAs exert extensive cardiac effects. The development of commercial solutions of FO opens perspectives for therapeutic applications in patients with acute cardiac conditions.the 3 following hypotheses will be addressed in patients requiring cardiac surgery under cardiopulmonary bypass or after myocardial infarction:perioperative /post-PTCA intravenous fish oil modifies the composition of membrane phospholipids in platelets and cardiac cells, blunts the physiological response to cardiac surgery/myocardial infarction, and reduces the incidence of arrhythmias, and reduces the occurrence of systolic dysfunction.

DETAILED DESCRIPTION:
A. Randomized trial in 40 cardiac surgery patients Early rapid infusion of fish oil (3 times in 24 hours) in cardiac surgery patients.

B. Randomized trial 20 myocardial infarction patients (abandonned) Continuous infusion of the same dose over 24hrs in the myocardial infarction patients

Additional trial in healthy volunteers (investigating physiological changes after cardiac study):

-Open trial in 8 healthy lean volunteers to investigate the impact of the same 0.6 g/kg FO dose IV (Week 1: 3hrs), and then orally on week 2, on platelet n-3 PUFA incorporation, platelet function, heart rate and peak flow response to stress test.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease requiring elective surgical repair under cardiopulmonary bypass
* Acute myocardial infarction requiring ICU management

Exclusion Criteria:

* Absence of consent
* Ventricular ejection fraction < 35%
* Beating heart surgery or emergency surgery
* Hypercholesterolemia > 5 mmol/l
* Thrombolysis
* Chronic steroid therapy
* Acute or chronic renal failure prior to surgery (plasma creatinine > 150 umol/l)
* Chronic coagulation disorder
* Premenopausal female
* Consumption of more than 3 times fish per week

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-01; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Incorporation of n-3 PUFA into platelet cell membrane and myocardial tissue | 48 hours
  The primary outcome is the determination of magnitude of the incorporation and the time required for incorporation of omega-3 fatty acid cell membrane composition after short intravenous infusions was unknown until the present study (HPLC determination of fatty acid membrane composition in all patients)

SECONDARY OUTCOMES:
Inflammatory and metabolic response | From operation to ICU discharge (maximum 28 days)
  cytokine determination, CRP, glucose control (blood levels and insulin requirements) in all patients
Global clinical outcome | From operation to hospital discharge (maximum 28 days)
  length of mechanical ventilation, length of ICU and hospital stay in all patients
Myocardial recovery after surgery | From operation to hospital discharge (maximum 28 days)
  Holter monitoring during cardiac surgery or for 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mette M Berger, MD, PhD, Study Director — Serviceof Adult Intensive Care, CHUV
Locations (2):
- Switzerland (2):
  - CHUV, Lausanne, Canton of Vaud
  - Service of Adult Intensive Care - CHUV, Lausanne, Canton of Vaud

REFERENCES:
- [Result] Berger MM, Delodder F, Liaudet L, Tozzi P, Schlaepfer J, Chiolero RL, Tappy L. Three short perioperative infusions of n-3 PUFAs reduce systemic inflammation induced by cardiopulmonary bypass surgery: a randomized controlled trial. Am J Clin Nutr. 2013 Feb;97(2):246-54. doi: 10.3945/ajcn.112.046573. Epub 2012 Dec 26. PMID 23269816
- [Derived] Delodder F, Tappy L, Liaudet L, Schneiter P, Perrudet C, Berger MM. Incorporation and washout of n-3 PUFA after high dose intravenous and oral supplementation in healthy volunteers. Clin Nutr. 2015 Jun;34(3):400-8. doi: 10.1016/j.clnu.2014.07.005. Epub 2014 Jul 15. PMID 25066733